CLINICAL TRIAL: NCT01075607
Title: The Comparison of Lymph Fluid and Blood From Metastatic and Non-metastatic Invasive Breast Cancer Patients for Identification of Novel Biomarkers
Brief Title: Lymph Fluid and Blood Collection for Identification of Novel Biomarkers
Status: Terminated | Type: Observational
Why Stopped: Halted prematurely due to lack of funding.
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 0911-04
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Adenocarcinoma of the Breast
Keywords: Lymph fluid collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to identify and validate metastasis protein markers in lymph collected from women with metastatic breast cancer. We will examine peripheral blood for the presence of these identified markers in order to develop a user friendly clinical test to detect metastasis and to evaluate response to therapy.

DETAILED DESCRIPTION:
The goal of the study is to identify node-negative breast cancer patients who are unlikely to benefit from adjuvant chemotherapy, thus saving them from the adverse effects of unnecessary treatment. We propose to identify and validate protein markers that can determine breast cancer recurrence and metastasis, based on an approach our group has recently found highly promising for biomarker discovery.

The objective of our research is to identify and validate metastasis protein markers in lymph collected from vessels exiting from the primary tumor and prior to their entry into sentinel lymph node in women with metastatic breast cancer. Realizing that this novel procedure cannot be adopted for routine clinical use, we will examine the peripheral blood for the presence of these identified markers in order to develop a user friendly clinical test to detect metastasis and to evaluate response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women, age greater than or equal to 18, with histologically and/or cytologically confirmed diagnosis of adenocarcinoma of the breast with metastatic (node positive) and/or non-metastatic (node negative) breast cancer.
* No prior chemotherapy treatment.
* Women, age greater than or equal to 18, with carcinoma in situ that opted for mastectomy.
* Able to provide informed consent and HIPAA authorization.

Exclusion Criteria:

* Hormone therapy in the past six months. Birth control pill use is allowed.
* History of radiation therapy to the chest.
* Previous or current use of aromatase inhibitor (AI) or Selective Estrogen Receptor Modulator (SERM) medication.
* History of chemotherapy for breast or other cancers.
* Pregnant or breast-feeding.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with adenocarcinoma of the breast - no prior chemotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2020-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Identification and Validation of Metastasis Protein Markers | Every 6 mo. for 5 years
  Lymph fluid collected at surgery; blood collected at surgery and then every 6 months for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Monet Bowling, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States